CLINICAL TRIAL: NCT04883437
Title: An Open-Label Phase 2 Trial of Acalabrutinib Plus Obinutuzumab in Patients With Untreated, Low Tumor Burden Follicular Lymphoma and Other Indolent Non-Hodgkin Lymphomas
Brief Title: Acalabrutinib and Obinutuzumab for the Treatment of Previously Untreated Follicular Lymphoma or Other Indolent Non-Hodgkin Lymphomas
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: AstraZeneca (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jonathon Cohen, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002247; NCI-2021-00894 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00002247; WINSHIP5186-20 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2021-05-07; First posted 2021-05-12 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Grade 1 Follicular Lymphoma; Grade 2 Follicular Lymphoma; Grade 3a Follicular Lymphoma; Indolent Non-Hodgkin Lymphoma; Lymphoplasmacytic Lymphoma; Lymphoproliferative Disorder; Mantle Cell Lymphoma; Marginal Zone Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Lymphoproliferative Disorders; Lymphoma, Mantle-Cell | interventions — acalabrutinib; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (acalabrutinib, obinutuzumab) (Experimental): INDUCTION PHASE: Patients receive acalabrutinib PO BID on days 1-28. Patients also receive obinutuzumab IV on days 1, 8, and 15 of cycle 3, then on day 1 of cycles 4-8. Treatments repeat every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  FOLLOW-UP PHASE: After cycle 12, patients who are in CR are randomized to either discontinue acalabrutinib or to continue acalabrutinib monotherapy in the absence of disease progression or unacceptable toxicity. Patients with PR or SD after cycle 12 continue acalabrutinib monotherapy in the absence of disease progression or unacceptable toxicity. Patients with disease progression after cycle 12 discontinue study treatment. Patients with disease progression at any time prior to the conclusion of cycle 12 may continue study therapy if they are felt to be benefiting by the treating physician, but not past cycle 12.
  Interventions: Drug: Acalabrutinib; Biological: Obinutuzumab; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Acalabrutinib — Given PO
  Other Names: ACP-196; Bruton Tyrosine Kinase Inhibitor ACP-196; Calquence
Biological: Obinutuzumab — Given IV
  Other Names: Anti-CD20 Monoclonal Antibody R7159; GA-101; GA101; Gazyva; huMAB(CD20); R7159; RO 5072759; RO-5072759; RO5072759
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies the effect of acalabrutinib and obinutuzumab in treating patients with follicular lymphoma or other indolent non-Hodgkin lymphoma for which the patient has not received treatment in the past (previously untreated). Acalabrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Immunotherapy with obinutuzumab may induce changes in body's immune system and may interfere with the ability of cancer cells to grow and spread. Giving acalabrutinib and obinutuzumab may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if treatment acalabrutinib and obinutuzumab is effective in patients with untreated, low tumor burden follicular lymphoma and other indolent non-Hodgkin lymphomas (NHLs).

SECONDARY OBJECTIVES:

I. Determine the complete response (CR) rate for single agent acalabrutinib at the end of a single-agent run-in for patients with untreated low tumor burden follicular lymphoma (FL).

II. Determine tolerability of acalabrutinib and obinutuzumab via assessment of patient-reported outcomes and conventional assessments.

III. Assess duration of response and long-term outcomes including progression-free survival.

IV. Assess the impact of early treatment with this regimen on health-related quality of life.

TERTIARY/EXPLORATORY OBJECTIVES:

I. Evaluate the impact of treatment discontinuation in patients who have achieved a complete response at the end of the induction phase.

II. To assess the safety and efficacy of acalabrutinib and obinutuzumab in other subtypes of indolent NHL.

OUTLINE:

INDUCTION PHASE: Patients receive acalabrutinib orally (PO) twice daily (BID) on days 1-28. Patients also receive obinutuzumab intravenously (IV) on days 1, 8, and 15 of cycle 3, then on day 1 of cycles 4-8. Treatments repeat every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.

FOLLOW-UP PHASE: After cycle 12, patients who are in CR are randomized to either discontinue acalabrutinib or to continue acalabrutinib monotherapy in the absence of disease progression or unacceptable toxicity. Patients with partial response (PR) or stable disease (SD) after cycle 12 continue acalabrutinib monotherapy in the absence of disease progression or unacceptable toxicity. Patients with disease progression after cycle 12 discontinue study treatment. Patients with disease progression at any time prior to the conclusion of cycle 12 may continue study therapy if they are felt to be benefiting by the treating physician, but not past cycle 12.

After completion of study treatment, patients are followed up at 30 days, every 12 weeks for 1 year, then every 6 months until disease progression or next anti-lymphoma treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men and women >= 18 years of age
* Patients will need to have one of the following clinical scenarios:

  * Previously untreated follicular lymphoma grade 1-3a with low tumor burden by Groupe d'Etude des Lymphomes Folliculaires (GELF) criteria
  * Previously untreated follicular lymphoma grade 1-3a with high tumor burden by GELF criteria but who are unable or unwilling to receive standard front-line treatment approaches
  * Previously untreated marginal zone lymphoma, lymphoplasmacytic lymphoma, or any other indolent B-cell lymphoproliferative disorder with low tumor burden by GELF criteria or who are unable/unwilling to receive more intensive front-line treatment
  * Previously untreated mantle cell lymphoma who would otherwise be appropriate candidates for watchful waiting OR who have symptomatic disease but are not candidates for or decline standard induction approaches
* Patients with previously untreated low tumor burden FL (criterion above) must have measurable and/or assessable disease defined as at least one involved lymph node or extranodal disease site that measures >= 1.5cm in greatest diameter
* Patients who meet inclusion criteria above are eligible as long as they meet one of the following criteria for measurable/assessable disease:

  * At least one involved lymph node or extranodal disease site measuring > 1.5cm in greatest diameter
  * Pathologically-confirmed bone marrow or peripheral blood involvement that can be reassessed for response
  * Pathologically confirmed splenic or extranodal involvement with at least one known site of disease remaining after diagnostic biopsy that can be reassessed (i.e., patients with splenic marginal zone lymphoma who complete splenectomy and have no other detectable disease would not be eligible)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Woman of childbearing potential (WOCBP) and men enrolled on this protocol must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry for the duration of study participation, and for at least 2 days after the last dose of acalabrutinib or 18 months after the last dose of obinutuzumab, whichever is longer. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Women of childbearing potential must have a negative serum or urine pregnancy test prior to starting therapy
* Willing and able to participate in all required evaluations and procedures in this study protocol
* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information

Exclusion Criteria:

* The presence or history of histologically transformed or co-existing high-grade or aggressive non-Hodgkin lymphoma
* Confirmed active or prior central nervous system disease
* Prior receipt of lymphoma-directed therapy or prior antibody-based therapy (except for anti-microbial therapy for infection-associated marginal zone lymphoma such as hepatitis C or H pylori)

  * A short course of steroids is permitted for patients aside from those in the low tumor burden FL cohort. This course may be no more than 14 days and steroids must be discontinued (or tapered to =< 10mg prednisone or equivalent) no later than 3 days after initiation of study treatment. Patients in the low tumor burden FL cohort may not receive corticosteroids as an anti-lymphoma therapy at any time before starting treatment
* Prior malignancy (or any other malignancy requiring active treatment), except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer from which the subject has been disease free for >= 2 years or which will not limit survival to < 5 years
* Clinically significant cardiovascular disease such as symptomatic ventricular arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification. Note: Subjects with controlled, asymptomatic atrial fibrillation can enroll on study if deemed appropriate by the investigator
* Has difficulty with or is unable to swallow oral medication, or has significant gastrointestinal disease that would limit absorption of oral medication
* Known history of human immunodeficiency (HIV) or any active significant infection (e.g., bacterial, viral, or fungal) within 14 days of cycle 1. Patients with uncomplicated viral or bacterial infections that are being managed with oral antibiotics and/or supportive care alone are eligible
* Known history of hypersensitivity or anaphylaxis to study drug(s) including active product or excipient components
* Active bleeding or history of bleeding diathesis (e.g., hemophilia or von Willebrand disease)
* Uncontrolled AIHA (autoimmune hemolytic anemia) or ITP (idiopathic thrombocytopenic purpura)
* Presence of a gastrointestinal ulcer diagnosed by endoscopy within 3 months before screening
* Requires treatment with a strong cytochrome P450 3A4 (CYP3A4) inhibitor/inducer
* Requires or receiving anticoagulation with warfarin or equivalent vitamin K antagonists
* Requires treatment with proton pump inhibitors (e.g, omeprazole, esomeprazole, lansoprazole, dexlansoprazole, rabeprazole, or pantoprazole). Note: Subjects receiving proton pump inhibitors who switch to H2-receptor antagonists or antacids are eligible for enrollment to this study
* History of significant cerebrovascular disease/event, including stroke or intracranial hemorrhage, within 6 months before the first dose of study drug. Patients with a transient ischemic attack which has resolved and for which there are no ongoing symptoms are eligible
* Major surgical procedure within 28 days of first dose of study drug (not including a diagnostic procedure to make the lymphoma diagnosis). Note: If a subject had major surgery, they must have recovered adequately from any toxicity and/or complications from the intervention before the first dose of study drug
* Hepatitis B or C serologic status: subjects who are hepatitis B core antibody (anti-HBc) positive and who are hepatitis B surface antigen (HBsAg) negative will need to have a negative polymerase chain reaction (PCR) and must be willing to undergo deoxyribonucleic acid (DNA) PCR testing during the study to be eligible. Those who are HBsAg positive or hepatitis B PCR positive will be excluded. Subjects who are hepatitis C antibody positive will need to have a negative PCR result to be eligible and have completed appropriate anti-viral treatment. Those who are hepatitis C PCR positive will be excluded. Anti-viral therapy for patients with hepatitis-C associated marginal zone lymphoma will not be considered a prior anti-lymphoma treatment
* Absolute neutrophil count (ANC) < 1,000/mcL
* Platelet count < 50,000/mcL (Unless felt to be related to underlying disease)
* Total bilirubin >= 1.5 x the upper limit of normal (ULN). Isolated bilirubin > 1.5 x ULN is permitted if the direct proportion is < 35%
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) > 2.5 x ULN
* Creatinine clearance =< 40 mL/min/1.73m^2
* Breastfeeding or pregnant
* Concurrent participation in another therapeutic clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2021-09-03 (Actual); Primary Completion 2026-09-23 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Complete response (CR) rate | Up to start of cycle 6 (each cycle = 28 days)
  Complete response rate will be calculated, and a 95% confidence interval will be estimated using the Clopper-Pearson method.
Incidence of grade 3+ adverse events | Up to 30 days post treatment
  Assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

SECONDARY OUTCOMES:
Overall response rate | Up to 3 years
  Overall response rate will be calculated, and a 95% confidence interval will be estimated using the Clopper-Pearson method.
CR rate for acalabrutinib monotherapy at end of single-agent run-in | Up to 3 years
  Will be calculated, and a 95% confidence interval will be estimated using the Clopper-Pearson method.
2-year progression free survival (PFS) | From first dose to documented disease progression, or death from any cause, whichever occurs first, assessed at 2 years
  PFS will be estimated using Kaplan-Meier methodology. Approximate 95% confidence intervals (CIs) for median PFS will be computed using the Brookmeyer and Crowley method.
Overall survival (OS) | From first dose to death from any cause, assessed up to 3 years
  Duration of OS will be estimated using Kaplan-Meier methodology. Approximate 95% CIs for median OS will computed using the Brookmeyer and Crowley method.
Duration of response (DOR) | From the first tumor assessment supports the response to the time of confirmed disease progression or death due to any cause, whichever occurs first, assessed up to 3 years
  DOR will be estimated using Kaplan-Meier method. Approximate 95% CIs for median DOR will be computed using the Brookmeyer and Crowley method.
Time to next anti-lymphoma treatment | From the end of induction visit up to and including the date of initiation of next treatment for any reason, assessed up to 3 years
  Time to next anti-lymphoma treatment is defined as the time from the end of induction visit up to and including the date of initiation of next treatment for any reason. This includes any chemotherapy, antibody therapy, oral therapy, and radiation therapy. Time to next anti-lymphoma treatment will be estimated using Kaplan-Meier methodology. Approximate 95% CIs for median time to next anti-lymphoma treatment will be computed using the Brookmeyer and Crowley method
Quality of life (QOL) assessments | Up to 3 years
  QOL measures from the Functional Assessment of Cancer Therapy General questionnaire obtained during treatment will be compared to the baseline values obtained at the screening visit using paired t-tests, McNemar's tests, or their nonparametric equivalents, where appropriate.
Patient-reported adverse events. | Up to 3 years
  Categorical Patient Reported Outcomes (PRO)-CTCAE variables will be summarized using frequencies and percentages, and numeric PRO-CTCAE variables will be summarized using mean, median, standard deviation, interquartile range (IQR), and range.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathon B Cohen, MD, MS, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia, United States

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-15): https://cdn.clinicaltrials.gov/large-docs/37/NCT04883437/Prot_SAP_000.pdf
  • Informed Consent Form (2025-07-22): https://cdn.clinicaltrials.gov/large-docs/37/NCT04883437/ICF_001.pdf